CLINICAL TRIAL: NCT05445193
Title: PEaters Choice™: Randomized Control Trial to Improve Picky Eating Behaviour Among Children Aged 3-5 Years
Brief Title: PEaters Choice™: Nutrition Intervention Module for Picky Eaters
Acronym: PEaters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Dr Nur Hana Hamzaid, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PEatersChoice_NUMas
Record Dates: First submitted 2022-06-22; First posted 2022-07-06 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Picky Eating
Keywords: picky eaters; food repertoire; children eating behaviour; nutrition intervention module
MeSH Terms: conditions — Food Fussiness

STUDY DESIGN:
Intervention Model Description: This study is single-blinded, with balance randomization (1:1) and parallel-group design. Dyads will be recruited from chosen nurseries and kindergartens. Following that, the dyads will be randomly assigned to either an intervention group or a controlled group by using Microsoft Excel Random Number Generator. Dyads will then fill out the sociodemographic information form, the Child Healthy Eating Knowledge Questionnaire, and the food intake form. The research team will also measure the children's weight and height using standard methods. Next, the nutritional status of each child is assessed by using WHO Anthro Software version 3.2.2.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Module PEaters Choice™ (Experimental): Using module that will be develop
  Interventions: Behavioral: PEaters Choice Module
- Standard nutrition information (No Intervention): No intervention done, just a standard information about nutrition.

INTERVENTIONS:
Behavioral: PEaters Choice Module — There will be nine sessions conducted throughout the intervention period, which include module activity, assessment sessions and follow-up sessions. This module will have four primary sub modules (SM): SM1- An overview of picky eaters, SM2-Healthy eating for children, SM3-Parental Strategies and SM4- Sensory perception.
  Arms: Module PEaters Choice™

SUMMARY:
Picky eaters (PE) are defined as individuals with a lack of diversity in food intake and fear of trying new foods which generally leads to malnutrition. Globally, between 20% to 55% of children worldwide are being reported as PE. Malaysia particularly has 31.8% PE children. To date, limited comprehensive modules on dietary recommendations are designed to help parents and/or primary healthcare workers to address this issue. This study is a single-blind randomized controlled trial to evaluate the effectiveness of PEaters Choice™ designed for PE children aged three to five years, with the objective to increase the food repertoire of the children. The PEaters Choice™ is a 12-week intervention program designed for mother, father or guardian-child dyads. The dyads will be divided into two groups; Intervention and Control Group. This trial will require each group to complete a list of commonly eaten foods, Child Eating Behavior Questionnaires, and a set of anthropometric data. Intervention groups will then follow three phases of the intervention program. This module suits primary healthcare settings, helping parents or guardians strategize meal planning, hence lowering the risk of malnutrition among PE children.

DETAILED DESCRIPTION:
The study will be conducted at the UKM Specialist Children's Hospital (HPKK UKM) in Kuala Lumpur to simulate real-life situations for this module. All briefings, therapies, and activities will be conducted in this setting. Considering several factors, especially subjects' commitment to attend the prescribed session, the selected area to participate in the study is a 5km radius from HPKK UKM.

The study information sheet and consent form are written in Malay, the Malaysian national language, and in the English language. The head researcher is responsible for the consent process and answering all relevant questions. However, other researchers will also assist in conveying this information from time to time. After the briefing session, mother, father or guardian will be given time to understand and ask any questions related to the study. If the parents or guardians feel it is necessary to take a longer time before making a decision, they may also take the study information form and consent form home.

Sample size calculation using the G-Power program (95% confidence interval, 80% power) found a minimum of 138 subjects required. The study sample was increased by 10%, considering the dropout factors to 154 subjects (77 people for each group).

The dyads who have consented to participate in the study will be placed in the same age nursery or kindergartens group and randomly selected to participate in intervention groups. Children in the same nursery/kindergarten will receive the same intervention. As the intervention will be conducted by the researcher, the dyads will not be informed (blinded) of their type of intervention.

The research team will manage all data. Data will be entered into the SPSS program by the researcher and reviewed by the head researcher. Questionable data will be confirmed with original forms or relevant sources. Outlier data that is deemed unreasonable will be removed and marked as missing.

Most of the questionnaires will be filled out by mothers, fathers or guardians, in ensuring they understand the questions correctly. To avoid data loss, each form will be carefully reviewed once completed by mothers, fathers or guardians. Weighing scales and stadiometers will always be calibrated using standard weights and rulers before weight and height measurements are taken. The head researcher will check 10% of the BMI calculation and nutritional status as a quality control measure.

Data will be analyzed using the SPSS program. Using mixed ANOVA, the investigators compared the list of foods eaten (food repertoire) before, during, and after the intervention between the two groups to evaluate the impact of the intervention. On the Child Eating Behavior Questionnaires, the comparison of eight primary constructs scores between the two groups was also accomplished with mixed ANOVA. A similar statistical analysis was used to assess the nutritional status of the intervention and control groups.

All data will be kept in a safe location that only the research team will have access to. Password protection will be implemented on all user computers. Once the data is no longer required for this study, it will be destroyed. After the trial ends, the data will be kept for at least three years. The trial data will be disposed of in compliance with the Malaysian Good Clinical Practice Guidelines 2018, which will be followed.

The procedure in this study will not involve any invasive process and provided only minimal risk to the subjects. Therefore, the subjects will continue participating in the study for 12 weeks. If any subject fails to attend two consecutive therapy/activity sessions and does not attend three sessions in total, the subject will be removed from the study. However, the final decision to discontinue the subject will be made after discussion with the research team members.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are between three and five years old
* Subjects had PE problems (screened using the CEBQ)

Exclusion Criteria:

* subject has clinical health problems such as autism, down syndrome, global developmental delay, dyslexia, or any health problem interfering with eating habits.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 154 (Estimated)
Dates: Start 2023-03 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change of food repertoire from baseline at sixth weeks | The list will be collected at the sixth weeks.
  List of food eaten by the subject
Change of food repertoire from baseline at 12th weeks | The list will be collected the 12th weeks.
  List of food eaten by the subject

SECONDARY OUTCOMES:
Change of children's eating behaviors (CEBQ) from baseline at sixth weeks | It will be collected at the sixth weeks
  CEBQ is an instrument used to identify eating behaviors for children. There are eight primary constructs: 1) food responsiveness 2) enjoyment of food 3) emotional-overeating 4) desire to drink 5) satiety responsiveness 6) slowness in eating 7) emotional under-eating 8) food fussiness. Each question must be answered using a Likert scale with a choice of 5 answers, namely never (1), rarely (2), sometimes (3), often (4), and always (5). A high average score for each construct indicates a high intensity for the behaviour.
Change of children's eating behaviors (CEBQ) from baseline at 12th weeks | It will be collected at the 12th weeks
  CEBQ is an instrument used to identify eating behaviors for children. There are eight primary constructs: 1) food responsiveness 2) enjoyment of food 3) emotional-overeating 4) desire to drink 5) satiety responsiveness 6) slowness in eating 7) emotional under-eating 8) food fussiness. Each question must be answered using a Likert scale with a choice of 5 answers, namely never (1), rarely (2), sometimes (3), often (4), and always (5). A high average score for each construct indicates a high intensity for the behaviour. The construct used in the CEBQ is food fussiness, with six questions to assess PE behaviour. Children were categorized as PE if they obtained a mean value of three and above
Change of weight-for-age (z-scores) from baseline at sixth weeks | It will be collected at the sixth weeks
  Weight and height will be collected and weight-for-age (z-scores) will be assessed through a WHO Anthro Software.
Change of weight-for-age (z-scores) from baseline at 12th weeks | It will be collected at the 12th weeks
  Weight and height will be collected and weight-for-age (z-scores) will be assessed through a WHO Anthro Software.
Change of height-for-age (z-scores) from baseline at sixth weeks | It will be collected at the sixth weeks
  Weight and height will be collected and height-for-age (z-scores) will be assessed through a WHO Anthro Software.
Change of height-for-age (z-scores) from baseline at 12th weeks | It will be collected at the 12th weeks
  Weight and height will be collected and height-for-age (z-scores) will be assessed through a WHO Anthro Software.
Change of weight-for-height (z-scores) from baseline at sixth weeks | It will be collected at the sixth weeks
  Weight and height will be collected and weight-for-height (z-scores) will be assessed through a WHO Anthro Software.
Change of weight-for-height (z-scores) from baseline at 12th weeks | It will be collected at the 12th weeks
  Weight and height will be collected and weight-for-height (z-scores) will be assessed through a WHO Anthro Software.
Change of BMI-for-age (z-scores) from baseline at sixth weeks | It will be collected at the sixth weeks
  Weight and height will be collected and Body Mass Index (BMI) is calculated from weight and height readings. Then, BMI-for-age will be assessed through a WHO Anthro Software.
Change of BMI-for-age (z-scores) from baseline at 12th weeks | It will be collected at the 12th weeks
  Weight and height will be collected and Body Mass Index (BMI) is calculated from weight and height readings. Then, BMI-for-age will be assessed through a WHO Anthro Software.

CONTACTS AND LOCATIONS:
Overall Officials: Nur Hana Hamzaid, Principal Investigator — National University of Malaysia
Locations (1):
- UKM Specialist Children's Hospital, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Only the research team and the Research Ethics Committee (REC), UKM can access this data. Data will be reported collectively without reference to individuals. Therefore subject identity and personal data will be kept confidential.

REFERENCES:
- [Background] Goh DY, Jacob A. Perception of picky eating among children in Singapore and its impact on caregivers: a questionnaire survey. Asia Pac Fam Med. 2012 Jul 20;11(1):5. doi: 10.1186/1447-056X-11-5. PMID 22816553
- [Background] Li Z, van der Horst K, Edelson-Fries LR, Yu K, You L, Zhang Y, Vinyes-Pares G, Wang P, Ma D, Yang X, Qin L, Wang J. Perceptions of food intake and weight status among parents of picky eating infants and toddlers in China: A cross-sectional study. Appetite. 2017 Jan 1;108:456-463. doi: 10.1016/j.appet.2016.11.009. Epub 2016 Nov 4. PMID 27825943
- [Background] Machado BC, Dias P, Lima VS, Campos J, Goncalves S. Prevalence and correlates of picky eating in preschool-aged children: A population-based study. Eat Behav. 2016 Aug;22:16-21. doi: 10.1016/j.eatbeh.2016.03.035. Epub 2016 Apr 5. PMID 27077700
- [Background] Mohd Hanapi, H. & Mohd Fahmi Teng, N. I. 2022. Picky Eating Behaviour and Nutritional Status of Preschool Children in Kuala Selangor, Malaysia. Mal J Med Health Sci 18(1): 145-150.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-06-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT05445193/Prot_SAP_ICF_000.pdf